**Official Title of Study:** Dissemination strategies and implementation outcomes of adolescent character strength interventions.

NCT Number: N/A

**Document Date:** 12<sup>th</sup> April 2022

#### INFORMED CONSENT

My name is Tom Osborn (Chief Executive Director of Shamiri Institute). I am conducting a study titled:

Dissemination strategies and implementation outcomes of adolescent character strength interventions.

## **Purpose of the Study**

The purpose of the study is to understand how to disseminate an intervention to improve the wellbeing, academic success, social support, and mental health of high school students in Kenya. You may remember that you participated in one of these programs around three years ago. This research will give us information on how to spread this intervention to other students in Kenya and sub-Saharan Africa.

#### Procedures to be followed

Participation in this study will require that I ask you some questions about your wellbeing, social support and mental health using a questionnaire four times, over the course of two months. We will also collect your academic scores from the school staff. This information will be obtained through questionnaires which you will fill out yourself. We may contact you in the future to complete further questionnaires. After the study is completed, identified data will be destroyed.

# Voluntarism

You have the right to refuse participation in this study. You will get the same services and care whether you agree to join the study or not and your decision will not change the care you will receive. Please remember the participation in this study is voluntarily. You may ask questions related to the study at any time.

You may refuse to respond to any questions, and you may stop an interview at any time. You may also stop being in the study at any time without any consequences to the services you receive here or any other organization now or in the future.

#### **Discomforts and Risks**

Some of the questions you will be asked are on intimate subjects and may be embarrassing or make you feel uncomfortable. Additionally, some questions on the questionnaires participants are asked to fill out may make participants uncomfortable or may ask for information which participants do not wish to share. If that is the case, you may refuse to answer these questions if you choose. You may also stop the questionnaire at any time.

Another risk is the risk of loss of time. You will spend approximately 1 hour per week for four weeks, and an additional 20 minutes after a month participating in this study.

Finally, there is some risk that participants may reveal things in the peer groups that cause others to think of them or treat them differently. This could be emotionally distressing to participants. If this occurs, peer group leaders will reach out to school administrators, their

supervisors, and study staff as appropriate. Furthermore, you can reach out to your group leader as a resource to support you if you deem necessary. Finally, participants are free to drop out of the study at any time if they are feeling uncomfortable.

#### **Benefits**

If you participate in this study you will help us to learn how to provide an effective intervention that could be used more broadly in Kenya and elsewhere in the world to improve adolescent academic performance, wellness and mental health. You may benefit from participating in our study in a variety of different ways. First, you may learn and reinforce important skills for your future. Furthermore, you may notice improvements in your wellbeing and in your academic functioning and grades. In addition, you may also feel that you have closer social ties to classmates because of the groups.

#### Reward

In addition to the aforementioned benefits, you will have the option to participate in raffles to win prizes such as t-shirts, school supplies, or 300 KES.

# **Confidentiality**

No information that reveals your identity will be released or published without your consent. The questionnaires will be completed in a private setting, on your own. The questionnaires will be kept in a locked cabinet for safe keeping. Everything will be kept private and only shared with the study team.

#### **Contact Information**

If you have questions about the study, call Mr.Tom Osborn +25470640811 or speak with a member of the study team in person.

However, if you have questions about your rights as a study participant: You may contact Kenyatta University Ethical Review Committee Secretariat on\_secretary.kuerc@ku.ac.ke.

## Participant's statement

The above information regarding my participation in the study is clear to me. The study has been explained to me and I have been given a chance to ask questions and my questions have been answered to my satisfaction. My participation in this study is voluntary. I understand that my records will be kept private and that I can leave the study at any time

| Name of Participant: | |
|---|---|
| Signature or Thumbprint | Date |
| Name of Representative/Witness (where necessary) | ) Relationship to Subject |
| Investigators statement | |
| I, the undersigned, have explained to the volum procedures to be followed in the study and the risks | |
| Name of Interviewer | |
| Signature | Date |
| Signature | Date |

#### INFORMED ASSENT FOR CHILDREN

**Project Title:** Dissemination strategies and implementation outcomes of adolescent character strength interventions.

Protocol Number: PKU/2456/E1587

## **Research Investigators:**

Tom L. Osborn, Project Co-Director, affiliated to Shamiri Institute

Ms. Katherine E. Venturo - Conerly, Project Co-Director, Harvard University, and Shamiri Institute

Dr. Christine M. Wasanga, Project Co-Investigator, Kenyatta University

Dr. John R. Weisz, Project Co-Investigator, Harvard University

Dr. Eve Puffer, Project Co-Investigator, Duke University

Dr. David Ndetei, Project Co-Investigator, Africa Mental Health Research and Training Foundation

Dr. Thomas Rusch, Project Co-Investigator, WU Vienna University of Economics and Business

The investigators named above are doing a research project.

## These are the things we want you to know about research project:

We are asking you to be in a research study. Research is a way to test new ideas. Research helps us learn new things.

Whether or not to be in this research is your choice. You can say Yes or No. Whatever you decide is OK.

#### What is the study about?

The purpose of the study is to provide evidence for an intervention which has been shown to improve the wellbeing, academic success, social support, and mental health of high school students in Nairobi, Kiambu and Makueni and to contribute to research to better a) understand the psychosocial needs of and b) serve at-risk adolescents in Kenya. The significance of this study is that it will help us understand how to give a brief, positive-psychology focused intervention that is delivered by lay-providers in schools to a larger number of adolescents in sub-Saharan Africa.

# Why am I being asked to be in this research study?

This research will help to increase knowledge of ways to serve and improve the health outcomes of adolescents in Kenya and other countries in sub-Saharan Africa. You are being asked to be in the study because you possess the characteristics that were required for the study participants. You are a high school student and as we cannot visit all the high schools in Kenya. Therefore, you are representing many other students who we will not be able to reach.

#### What will happen during this study?

If you agree to be in this study, you will be divided into groups. All the groups will be taught cognitive and behavioral skills and information about psychology. You will be randomized to different group leaders. Groups will meet for one hour for four weeks. You will be asked to fill out questionnaires four weeks after the discussion groups are over. These sessions will be audio-recorded. We may contact you in the future to complete further questionnaires. After the study is completed, identified data will be destroyed.

Groups will meet for at least one hour for four weeks. You will be asked to fill out questionnaires for up to four weeks after the discussion groups are over. These sessions will be audio-recorded. We may contact you in the future to complete further questionnaires. After the study is completed, identified data will be destroyed.

# Will the study hurt/risks?

It is extremely unlikely that you will be hurt or put at risk by participating in the study. With that said, discussions in the groups may sometimes make you feel uncomfortable. Additionally, some questions on the questionnaires that you are asked to fill out may make you uncomfortable or may ask for information which you do not wish to share. If that is the case, you may refuse to answer the question or choose to leave the study.

Another possible risk is the risk of loss of time. You will spend approximately 1 hour per week for four weeks participating in this study. We expect that the benefits to participant wellbeing and academic performance may outweigh this risk. We will also ensure that you will not miss any class time because of the study.

Finally, there is some risk that you may reveal things in the groups that cause others to think of you or treat you differently. This may cause you to worry and become anxious. If this occurs, peer group leaders will reach out to school administrators, their supervisors, or a member of the study team that is a professional psychologist as appropriate and defer to your school's standard procedures. Furthermore, you should feel free to reach out to your group leader if you think it is necessary. Finally, participants are free to drop out of the study at any time if they are feeling uncomfortable.

#### What else should I know about the study?

If you feel sick or afraid that something is wrong with you, speak to your group leader who will know what to do. You do not have to answer any questions that are asked of you.

# What are the good things /benefits that might happen?

During each session as an incentive to attend, a student present will be selected at random through a lottery to receive a small prize (i.e., water bottle, T-shirt or KES 300).

While we cannot guarantee benefits to participants, you may benefit from participating in our study in a variety of different ways. First, you may notice improvements in your wellbeing and in your academic functioning and grades. You may learn and reinforce important skills for the future. In addition, you may also feel that you have closer social ties to your classmates in the groups. More broadly, if successful, the intervention could be used throughout in Kenya and elsewhere to improve students' mental health and academic success.

## What if I don't want to be in this study?

Participation in this research is voluntary, and you can leave the research at any time it will not be held against you. You may ask questions related to the study at any time. You may refuse to respond to any questions, and you may stop an interview at any time.

# Who should I ask if I have any questions?

If you have questions about the study, you or your parents can call Tom Osborn at 0756121145. However, if you have questions about your rights as a study participant: You may contact Kenyatta University Ethical Review Committee Secretariat on <a href="mailto:chairman.kuerc@ku.ac.ke">chairman.kuerc@ku.ac.ke</a>, or, <a href="mailto:secretary.kuerc@ku.ac.ke">secretary.kuerc@ku.ac.ke</a>, or, <a href="mailto:secretary.kuerc@ku.ac.ke">secretary.kuerc@ku.ac.ke</a>, or,

# Do I have to be in the study?

No, you do not have to be in the study. Even if you say yes now, you can change your mind later. It is up to you. No one will be mad at you if you don't want to do this.

# **Signatures**

Before deciding if you want to be in the study, ask any questions you have. You can also ask questions during the time you are in the study.

If you sign your name or put a mark below, it means that you agree to take part in this research study.

| Your Name (Printed) | Age |
|---------------------------------------|-----------|
| Your Signature | Date |
| Signature of Person Obtaining Consent | Date |
| Signature of Witness | —————Date |